CLINICAL TRIAL: NCT00869128
Title: A Randomized Double-Blind, Crossover Study Comparing the Efficacy of Prolonged-Release Melatonin Versus Placebo in a 3 Week Treatment of Diabetic Patients Suffering From Insomnia
Brief Title: A Study of the Efficacy of Prolonged-Release Melatonin Versus Placebo in Diabetic Patients Suffering From Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Dr. Doron Garfinkel, Shoham Geriatric Medical Center,Pardes Hana 37000, Israel
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Neu951005
Record Dates: First submitted 2008-12-08; First posted 2009-03-25 (Estimated); Results first posted 2009-03-25 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes Mellitus, Type 2; Insomnia
Keywords: melatonin; insomnia; diabetes; sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Initiation and Maintenance Disorders; Diabetes Mellitus | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo First (Other): Subjects were treated for 3 weeks with 1 tablet per night of Placebo and then with 2 mg melatonin (Circadin).
  Interventions: Drug: Circadin; Drug: Placebo
- Circadin first (Other): Subjects were treated for 3 weeks with 1 tablet per night of 2 mg melatonin (Circadin) and then with placebo.
  Interventions: Drug: Circadin; Drug: Placebo

INTERVENTIONS:
Drug: Circadin — 2 mg prolonged-release melatonin
  Other Names: Prolonged-release melatonin (2mg)
Drug: Placebo

SUMMARY:
Objective - Type 2 uncontrolled diabetic patients often have low endogenous melatonin and suffer from sleep disorders. The effect of a prolonged-release melatonin (PRM) formulation on glucose lipid metabolism and sleep is studied in type 2 diabetes patients with insomnia.

DETAILED DESCRIPTION:
Methods: In a randomized, double-blind, crossover study, the subjects were treated for 3 weeks with 1 tablet per night of 2 mg prolonged-release melatonin or placebo, with one week washout period in between. Sleep was objectively monitored by wrist actigraphy. Fasting glucose, fructosamine, insulin, C-peptide, triglycerides, cholesterol (total, HDL and LDL) and some antioxidants were assessed at baseline and end of each period.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with proven presence of the disease who complained of insomnia.

Exclusion Criteria:

* Patients with liver or renal problems (serum creatinine above 1.5 mg/dL).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1995-11; Primary Completion 1997-03 (Actual); Study Completion 1997-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doron Garfinkel, MD, Principal Investigator — Department of Evaluation & Rehabilitation and Palliative Unit, Shoham Geriatric Medical Center, Pardes Hana, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 independently living patients who complained of insomnia and suffered from type 2 diabetes (16 treated with oral hypoglycemic agents and 20 on insulin) entered the study.
Pre-assignment Details: Patients with liver or renal disease (serum creatinine 1.5 mg/dL or higher) were excluded. All 36 patients were randomized and all concluded the crossover randomized and extension parts of the study.
Groups:
- Circadin First: Subjects were treated for 3 weeks with 1 tablet per night of Circadin 2mg and then with Placebo.
Period: Overall Study
Arm/Group | Placebo First | Circadin First
Started | 18 | 18
Completed | 12 | 12
Not Completed | 6 | 6
Not completed — lack of Compliance | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Subjects were treated for 3 weeks with 1 tablet per night of Placebo or Circadin and then 3 weeks of Circadin or Placebo, respectively.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 11
Region of Enrollment [Number; unit: participants]
  Israel | 36

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency
Description: Sleep efficiency is the percentage of time patients were asleep while in bed as scored by the actigraphic sleep algorithm assessed in the 3 consecutive last nights of each period
Time Frame: 3 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: Percentage of time asleep
Groups:
- Placebo: Subjects were treated for 3 weeks with 1 tablet per night of Placebo
- Circadin: Subjects were treated for 3 weeks with 1 tablet per night of Circadin 2mg
Arm/Group | Placebo | Circadin
Number analyzed (Participants) | 24 | 24
Percentage of time asleep | 79.5 (9.6) | 83.1 (11.3)
Statistical Analysis 1: Comparison: Placebo vs Circadin; ANOVA, The effect of Circadin was checked by means of 2 x 2 mixed design analysis of variance for repeated measurement; Test type: Superiority or Other; p = 0.04, ANOVA; The effect of Circadin was checked by means of 2 x 2 mixed design analysis of variance for repeated measurement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No